CLINICAL TRIAL: NCT01646866
Title: Early Detection of Autism Spectrum Disorder in Children
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: IntegraGen SA (Industry)
Responsible Party: Principal Investigator, Rolanda Gott, Assoc. Professor of Pediatrics, Professor of Pediatrics, St. Louis University
Other Study IDs: 15861
Record Dates: First submitted 2012-05-17; First posted 2012-07-20 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; siblings; genetic test; screening
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Siblings of Children with Autism Spectrum Disorders: This group is comprised of 6-12 month old siblings of a child with an expert clinical diagnosis of autism spectrum disorders.

SUMMARY:
Rationale: Autism Spectrum Disorder (ASD) is defined by deficits in social interaction and communication identified before the age of 3 years. Modified Checklist for Autism in Toddlers (M-CHAT) is a sensitive tool for ASD screening in children 16-23 months. A limited number of studies with a small number of patients have documented the developmental profile of children with ASD during infancy. Retrospective evaluations of videotaped behavior of children with ASD at 8 months and at 12 months identified early signs of ASD. A few studies found early signs of ASD during infancy in siblings of autistic children. Data documenting the age of onset and regression in ASD is controversial and limited. No large prospective studies documented the specific developmental profile of children with ASD starting at 6 months of age. Defining a specific autistic pattern on a developmental screening test could help identify infants at risk for ASD and improve their outcome through earlier diagnosis and treatment. More recently, genetic tests have been shown to aid in early identification of ASD which facilitates earlier intervention. Genetic testing among siblings of children with autism can aid in identification of autism or other related disorders in the siblings.

PURPOSE: The purpose of this study is to learn about the early signs of autism in siblings of children with autism spectrum disorders.

* The investigators will enroll siblings of children with ASD. Those siblings who completed the Red Flags for Communication scale (RFC) at 6 months and/or at 12 months and failed the RFC at 12 months will be given a genetic screening test.
* It is the investigators goal to define a specific autistic pattern on a developmental screening test that could help identify sibling infants at risk for ASD and improve their outcome through earlier diagnosis and treatment and to evaluate if the results of the clinical screening test will correlate with the results of the genetic screening test.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be a sibling of a child with a previous expert clinical diagnosis of Autism Spectrum Disorder.
* Subjects will be included for the genetic test if he/she meets the following criteria:

  * At 12 months of age he/she failed two or more items on the RFC with at least one failed critical item
  * They have no significant known hearing, vision or motor impairment that will impact on their ability to perform on developmental assessments

Exclusion Criteria:

* Those children who do not meet the inclusion criteria
* Those who do not speak English will be excluded from this study.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Biological siblings of children with a previous expert clinical diagnosis of Autism Spectrum Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Children with a High Risk Genetic Score on the ARISK Genetic Test who have a Diagnosis of Autism Spectrum Disorders (ASD) at 24 Months | 2 years

SECONDARY OUTCOMES:
Percentage of Children who failed the Red Flags for Communication (RFC) Scale at 12 months who have a Diagnosis of ASD at 24 months | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rolanda Gott, MD, Principal Investigator — St. Louis University
Locations (1):
- Knights of Columbus Developmental Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Robins DL, Fein D, Barton ML, Green JA. The Modified Checklist for Autism in Toddlers: an initial study investigating the early detection of autism and pervasive developmental disorders. J Autism Dev Disord. 2001 Apr;31(2):131-44. doi: 10.1023/a:1010738829569. PMID 11450812
- [Background] Osterling J, Dawson G. Early recognition of children with autism: a study of first birthday home videotapes. J Autism Dev Disord. 1994 Jun;24(3):247-57. doi: 10.1007/BF02172225. PMID 8050980
- [Background] Baranek GT. Autism during infancy: a retrospective video analysis of sensory-motor and social behaviors at 9-12 months of age. J Autism Dev Disord. 1999 Jun;29(3):213-24. doi: 10.1023/a:1023080005650. PMID 10425584
- [Background] Werner E, Dawson G, Osterling J, Dinno N. Brief report: Recognition of autism spectrum disorder before one year of age: a retrospective study based on home videotapes. J Autism Dev Disord. 2000 Apr;30(2):157-62. doi: 10.1023/a:1005463707029. No abstract available. PMID 10832780
- [Background] Osterling JA, Dawson G, Munson JA. Early recognition of 1-year-old infants with autism spectrum disorder versus mental retardation. Dev Psychopathol. 2002 Spring;14(2):239-51. doi: 10.1017/s0954579402002031. PMID 12030690
- [Background] Tuchman RF, Rapin I. Regression in pervasive developmental disorders: seizures and epileptiform electroencephalogram correlates. Pediatrics. 1997 Apr;99(4):560-6. doi: 10.1542/peds.99.4.560. PMID 9093299
- [Background] Goldberg WA, Osann K, Filipek PA, Laulhere T, Jarvis K, Modahl C, Flodman P, Spence MA. Language and other regression: assessment and timing. J Autism Dev Disord. 2003 Dec;33(6):607-16. doi: 10.1023/b:jadd.0000005998.47370.ef. PMID 14714930
- [Background] Lord C, Shulman C, DiLavore P. Regression and word loss in autistic spectrum disorders. J Child Psychol Psychiatry. 2004 Jul;45(5):936-55. doi: 10.1111/j.1469-7610.2004.t01-1-00287.x. PMID 15225337
- [Background] Rogers SJ. Developmental regression in autism spectrum disorders. Ment Retard Dev Disabil Res Rev. 2004;10(2):139-43. doi: 10.1002/mrdd.20027. PMID 15362172
- [Background] Siperstein R, Volkmar F. Brief report: parental reporting of regression in children with pervasive developmental disorders. J Autism Dev Disord. 2004 Dec;34(6):731-4. doi: 10.1007/s10803-004-5294-y. PMID 15679193
- [Background] Stone WL, McMahon CR, Yoder PJ, Walden TA. Early social-communicative and cognitive development of younger siblings of children with autism spectrum disorders. Arch Pediatr Adolesc Med. 2007 Apr;161(4):384-90. doi: 10.1001/archpedi.161.4.384. PMID 17404136
- [Background] Nadig AS, Ozonoff S, Young GS, Rozga A, Sigman M, Rogers SJ. A prospective study of response to name in infants at risk for autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):378-83. doi: 10.1001/archpedi.161.4.378. PMID 17404135
- [Background] Carayol J, Schellenberg GD, Dombroski B, Genin E, Rousseau F, Dawson G. Autism risk assessment in siblings of affected children using sex-specific genetic scores. Mol Autism. 2011 Oct 21;2(1):17. doi: 10.1186/2040-2392-2-17. PMID 22017886